CLINICAL TRIAL: NCT00202436
Title: Therapeutic Erythrocytapheresis as Treatment for Hemochromatosis Patients.
Brief Title: Haemochromatosis:Phlebotomy Versus Erythrocytapheresis Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Maastricht University Medical Center (Other); Atrium Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Dr.Wim de Kort PhD, Sanquin Blood Bank South-east
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPO-C- 03-006
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Hemochromatosis
MeSH Terms: conditions — Hemochromatosis | interventions — Phlebotomy; Bloodletting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Phlebotomy
  Interventions: Procedure: Phlebotomy; Procedure: Erythrocytapheresis
- 2 (Active Comparator): Erythrocytapheresis
  Interventions: Procedure: Phlebotomy; Procedure: Erythrocytapheresis

INTERVENTIONS:
Procedure: Phlebotomy — Removal of 500 ml whole blood
  Other Names: Bloodletting
Procedure: Erythrocytapheresis — machinal removal of erythrocytes
  Other Names: Therapeutic erythrocytapheresis

SUMMARY:
In this project we plan to evaluate the effectiveness of erythrocytapheresis against phlebotomy, both regarding the impact on the reduction in iron overload as well as reduction in patient "burden". Aspects of cost effectiveness will be included in the final analysis. Results of the study would allow decision-making based on Evidence Based Medicine on the "best" therapeutic options available for newly-diagnosed as well as existing primary hemochromatosis patients.

DETAILED DESCRIPTION:
In this project we plan to evaluate the effectiveness of erythrocytapheresis against phlebotomy, both regarding the impact on the reduction in iron overload as well as reduction in patient "burden". Aspects of cost effectiveness will be included in the final analysis. The results of the study would allow decision-making based on Evidence Based Medicine on the "best" therapeutic options available for newly-diagnosed as well as existing primary hemochromatosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary haemochromatosis patients

Exclusion Criteria:

* Malignancies, severe arrhythmias, congestive heart failure and/or recent angina, severe liver disease, epileptic seizures preceding in last 3 months before planned treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Treatment duration and number of treatments | Ferritine value 50 microgr/l

SECONDARY OUTCOMES:
Decline in hemoglobin levels, restitution in liver functions, patient discomfort en costs | Ferritine value 50microgr/l

CONTACTS AND LOCATIONS:
Overall Officials: Eva Rombout, MD, Principal Investigator — Sanquin Research and Blood Bank Divisions
Locations (1):
- Sanquin Blood Bank Southeast Region, Maastricht, Netherlands

REFERENCES:
- [Derived] Rombout-Sestrienkova E, Winkens B, van Kraaij M, van Deursen CTBM, Janssen MCH, Rennings AMJ, Evers D, Kerkhoffs JL, Masclee A, Koek GH. A predictive model for estimating the number of erythrocytapheresis or phlebotomy treatments for patients with naive hereditary hemochromatosis. J Clin Apher. 2021 Jun;36(3):340-347. doi: 10.1002/jca.21867. Epub 2020 Dec 24. PMID 33368569
- [Derived] Rombout-Sestrienkova E, Nieman FH, Essers BA, van Noord PA, Janssen MC, van Deursen CT, Bos LP, Rombout F, van den Braak R, de Leeuw PW, Koek GH. Erythrocytapheresis versus phlebotomy in the initial treatment of HFE hemochromatosis patients: results from a randomized trial. Transfusion. 2012 Mar;52(3):470-7. doi: 10.1111/j.1537-2995.2011.03292.x. Epub 2011 Aug 16. PMID 21848963